CLINICAL TRIAL: NCT02095587
Title: A Phase 1, Open-Label, Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Single Dose of Duvelisib in Subjects With Chronic Hepatic Impairment Compared to Healthy Subjects
Brief Title: Duvelisib in Hepatically Impaired Subjects Compared to Healthy Subjects
Acronym: IPI-145-14
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IPI-145-14
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Impairment
Keywords: Phase 1; hepatic impairment
MeSH Terms: interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: IPI-145
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: IPI-145
- Healthy Subjects (Experimental)
  Interventions: Drug: IPI-145
- Severe Hepatic Impairment (Experimental): Optional arm based on results from Arms 1, 2, and 3
  Interventions: Drug: IPI-145

INTERVENTIONS:
Drug: IPI-145 — 25 mg single oral capsule

SUMMARY:
To evaluate the pharmacokinetics, safety, and tolerability of IPI-145 when administered to subjects with chronic hepatic impairment and in matched healthy subjects.

DETAILED DESCRIPTION:
This is a nonrandomized, open-label, parallel-group, single oral dose study in subjects with chronic hepatic impairment and matched (age, sex, weight, BMI) healthy subjects. Subjects will be enrolled into 1 of 3 groups based on hepatic impairment grade: mild, moderate and normal hepatic function. An optional severe hepatic impairment group will enroll based on data from the mild and moderate hepatic impairment groups in comparison to matched healthy group. All subjects will receive a single oral dose of IPI-145 25 mg.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential between 18-70 years of age
* Body Mass Index (BMI): 18.0 - 38.0 kg/m2.
* Healthy subjects: in good health, determined by no clinically significant findings from clinical evaluations
* Hepatic impairment subjects: confirmed hepatic impairment >1 year with etiology of chronic alcoholism, chronic viral hepatitis (B or C), nonalcoholic steatohepatitis, autoimmune hepatitis, Wilson disease, alpha-1 antitrypsin deficiency, glycogen storage diseases, or galactosemia
* Provided written informed consent prior to any study specific procedures

Exclusion Criteria:

* Women of childbearing potential
* Hepatic impairment subjects: fluctuating or rapidly deteriorating hepatic function, acute hepatitis, variceal bleeding within 8 weeks of screening, a history of pancreatitis within 8 weeks of screening, evidence of hepatic encephalopathy > Grade 1, current unstable hematologic condition, and/or creatinine clearance < 60 mL/min
* Healthy subjects: positive screening test for hepatitis B surface antigen, or hepatitis C antibody
* ECG at screening or Day -1 showing QTcF ≥ 450 msec for healthy subjects or > 500 msec for hepatically impaired subjects
* Evidence of clinically significant medical conditions
* History of gastrointestinal disease or surgery that may affect drug absorption
* Positive or indeterminate QuantiFERON-TB Gold test at screening
* Any active infection at the time of screening or admission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of IPI-145 and its primary metabolite, IPI-656 | Open 72 hours
  PK parameters (AUC, Cmax and t1/2) of IPI-145 and its metabolite, IPI-656 Plasma concentrations of IPI-145 and its metabolite, IPI-656

SECONDARY OUTCOMES:
Incidence of adverse events following administration of IPI-145 | 10 days
  Safety Findings

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (1):
- Miami, Florida, United States